CLINICAL TRIAL: NCT07044960
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetic Profile of Single and Multiple Doses of KHN702 Tablets in Chinese Healthy Volunteers
Brief Title: A Phase 1 Study of KHN702 Tablets in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: KHN702-30101
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KHN702 tablet-Part I (Experimental): All participants will receive single dose of KHN702 tablet or placebo.
  Interventions: Drug: KHN702 tablet or placebo
- KHN702 tablet-Part II (Experimental): All participants will receive mutiple doses of KHN702 tablet or placebo.
  Interventions: Drug: KHN702 tablet or placebo

INTERVENTIONS:
Drug: KHN702 tablet or placebo — Subject will receive a single KHN702 tablet or matching placebo orally in fasted state.
  Arms: KHN702 tablet-Part I
Drug: KHN702 tablet or placebo — All participants will receive KHN702 tablet or matching placebo orally once a day for 7 days in fasted state.
  Arms: KHN702 tablet-Part II

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled study divided into a Single Ascending Dose (SAD) stage and a Multiple Ascending Dose (MAD) phase. The primary objective is to evaluate the safety and tolerability of KHN702 tablets in Chinese healthy volunteers（HVs).

DETAILED DESCRIPTION:
This study consists of two parts: Part 1-SAD phase and Part 2- MAD phase. There will be 7 cohorts in Part 1 and 3 cohorts in Part 2.

The SAD study will enroll approximately 54 HVs across 7 dose cohorts. All participants in Part 1 will be administered with a single oral dose of KHN702 or its matching placebo under fasted condition.

Approximately 30 HVs will be enrolled in the multiple ascending dose study. All participants in Part 2 will received KHN702 or placebo once daily for continuous 7 days (QD x 7d) in a double-blind manner.

The safety and tolerability will be evaluated by monitoring and assessment of AEs, clinical laboratory tests (hematology, urinalysis, biochemistry, coagulation, etc.), physical examination findings, etc.

ELIGIBILITY:
inclusion criteria:

1.Age: 18 to 45 years old (inclusive), Male or female. 2.Body weight: ≥ 50 kg for male and ≥ 45 kg for female, body mass index: 19~26 kg/m2 (inclusive).

3. Effective contraception measures and no sperm/egg donation plan from signing the informed consent to 3 months after last dose.

4.Fully understand the procedures and sigh the informed consent. exclusion criteria：

1. Have clinically significant medical history or clinical manifestations, including but not limited to the history of any clinically serious disease such as hematological system, circulatory system,digestive system, urinary system, respiratory system, central nervous system,immunology, endocrine system cardiovascular system, malignant tumors, metabolic abnormalities, or any other disease or physiological condition that may interfere with the results .
2. Subjects with clinically significant abnormalities in vital signs, physical examination, 12 lead electrocardiogram, laboratory examination, abdominal color Doppler ultrasound and chest X-ray during screening period, as determined by the investigator.
3. Dysphagia or history of gastrointestinal diseases, liver and kidney diseases that can affect the pharmacokinetic behavior of drugs as judged by the investigator.
4. Had surgery within 3 months before screening, or planned surgery during the study period, or had surgery that would affect drug absorption, distribution, metabolism, and excretion.
5. Allergic to the IMP or its excipients, or allergic to two or more other drugs, food and environment, or prone to skin rash, urticaria and other allergic symptoms.
6. Allergic to natural light / UV, or phototoxic reaction after previous use of specific drugs (such as fluoroquinolones and tetracyclines).
7. There are risk factors for cardiac disease, including but not limited to congenital long QT syndrome, torsade de pointes or torsade de pointes (such as hypokalemia, hypomagnesemia, family history of long QT syndrome). Currently, class IA [such as quinidine or procainamide] or class III [such as amiodarone or sotalol] antiarrhythmic drugs or other drugs known to affect QT interval are used. Or QTc interval (QTCF) corrected according to fridericia's criteria > 450 ms in males and > 470 ms in females at screening or other 12 lead ECG abnormalities with clinical significance.
8. Alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) and / or total bilirubin (TBIL), or serum creatinine (CR) exceeded the upper limit of normal at screening.
9. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and treponema pallidum antibody at Screening.
10. Systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg at screening.
11. Vaccinated within 30 days before screening.
12. Any drugs that affects the absorption, metabolism or elimination of the drug has been used within 30 days before administration.
13. Any drugs or health care products (including Chinese herbal medicine and vitamins) used within 14 days before the first administration of the study.
14. Have special requirements for diet and cannot comply with the unified diet.
15. Consumption of foods or juices containing alcohol or caffeine, or having strenuous exercise, or other factors affecting the absorption, distribution, metabolism, excretion of drugs with 48 hours before the first dose. Or disagree to stop drinking tea, coffee and / or caffeinated beverages and foods during the trial.
16. Average daily smoking of more than 5 cigarettes within the 3 months prior to screening or refuse to abstain from smoking during the trial.
17. A history of alcohol abuse or alcohol abuse within 6 months before screening (defined as an average intake of alcohol > 14 units per week, 1 unit ≈ 285 ml of beer with an alcohol content ≥ 3.5%, or 25 ml of spirits with an alcohol content ≥ 40%, or 85 ml of wines with an alcohol content ≥ 12%), or a positive alcohol test at the screening, or unable to abstain from alcohol during the trial.
18. Donation of blood or significant blood loss ≥ 400 mL in 3 month prior to screening.
19. Substance abuse-related disorder or a history of drug, or positive drug screen at screening and Day -1.
20. Positive pregnancy test, or lactating women.
21. Participate in other clinical trials within 3 months before screening (participation refers to receiving drug administration or device treatment for the trial).
22. Subjects with other factors deemed ineligible to participate in the trial by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-21 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AEs) | From screening to Day 4 for Part 1, and Day 10 for Part 2.
  Incidence and severity of adverse events (AEs), vital signs, physical examination, laboratory tests, electrocardiogram (ECG), etc.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.
Time to reach maximum observed concentration (Tmax) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.
Area under plasma concentration-time curve from zero to infinity (AUC0-inf) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.
Area under the plasma concentration-curve across the dosing interval (AUC0-tau) | Day 1 to Day 10.
  To characterise the steady state PK of KHN702 following oral multiple administration of KHN702.
Terminal elimination half-life (t1/2) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.
Apparent total body clearance (CL/F) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Part I: Day 1 to Day 4. Part II: Day 1 to Day 10.
  To characterise the single dose and steady state PK of KHN702 following oral administration of KHN702.

IPD SHARING:
Plan to Share IPD: Yes